CLINICAL TRIAL: NCT02666118
Title: Randomized Prospective Comparison of Analgesic Efficacy of Peripheral Nerve Blockade Performed Prior to Surgical Intervention Versus Following Surgical Shoulder Repair
Brief Title: Efficacy of Nerve Blockade Performed Prior to Surgical Intervention Versus Following Surgical Intervention
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2012-0486
Record Dates: First submitted 2016-01-26; First posted 2016-01-28 (Estimated); Last update posted 2024-04-02 (Actual); Status verified 2024-04

CONDITIONS: Pain; Shoulder Injury
Keywords: pain; pain management; shoulder repair; nerve blockade; regional anesthesia; pediatrics
MeSH Terms: conditions — Pain; Shoulder Injuries; Agnosia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor

ARMS (4):
- Preemptive Interscalene Block - Single Shot (Active Comparator)
  Interventions: Procedure: Preemptive Interscalene Block - Single Shot
- Postoperative Interscalene Block - Single Shot (Active Comparator)
  Interventions: Procedure: Postoperative Interscalene Block- Single Shot
- Preemptive Interscalene Block - Catheter (Active Comparator)
  Interventions: Procedure: Preemptive Interscalene Block - Catheter
- Postoperative Interscalene Block - Catheter (Active Comparator)
  Interventions: Procedure: Postoperative Interscalene Block - Catheter

INTERVENTIONS:
Procedure: Preemptive Interscalene Block - Single Shot — Interscalene brachial plexus blockade will be performed by the anesthesia team under ultrasound-guidance utilizing 1 ml/kg (to a maximum volume of 20 mls) of 0.2% ropivacaine without epinephrine. Regional anesthesia will be performed following the induction of anesthesia, but prior to the start of surgery. Anesthesia team members determined to be proficient in regional blockade, having performed a minimum of ten successful interscalene brachial plexus blocks previously, will be performing the regional blockade.
  Arms: Preemptive Interscalene Block - Single Shot
Procedure: Postoperative Interscalene Block- Single Shot — Interscalene brachial plexus blockade will be performed by the anesthesia team under ultrasound-guidance utilizing 1 ml/kg (to a maximum volume of 20 mls) of 0.2% ropivacaine without epinephrine. Regional anesthesia will be performed following the completion of surgery with the patient still under general anesthesia. Anesthesia team members determined to be proficient in regional blockade, having performed a minimum of ten successful interscalene brachial plexus blocks previously, will be performing the regional blockade.
  Arms: Postoperative Interscalene Block - Single Shot
Procedure: Preemptive Interscalene Block - Catheter — Interscalene brachial plexus blockade will be performed by the anesthesia team under ultrasound-guidance utilizing 1 ml/kg (to a maximum volume of 20 mls) of 0.2% ropivacaine without epinephrine. A continuous peripheral nerve catheter will then be placed under ultrasound-guidance for continuous infusion postoperatively. Regional anesthesia will be performed following the induction of anesthesia, but prior to the start of surgery. Anesthesia team members determined to be proficient in regional blockade, having performed a minimum of ten successful interscalene brachial plexus blocks previously, will be performing the regional blockade.
  Arms: Preemptive Interscalene Block - Catheter
Procedure: Postoperative Interscalene Block - Catheter — Interscalene brachial plexus blockade will be performed by the anesthesia team under ultrasound-guidance utilizing 1 ml/kg (to a maximum volume of 20 mls) of 0.2% ropivacaine without epinephrine. A continuous peripheral nerve catheter will then be placed under ultrasound-guidance for continuous infusion postoperatively. Regional anesthesia will be performed following the completion of surgery with the patient still under general anesthesia. Anesthesia team members determined to be proficient in regional blockade, having performed a minimum of ten successful interscalene brachial plexus blocks previously, will be performing the regional blockade.
  Arms: Postoperative Interscalene Block - Catheter

SUMMARY:
Nerve blocks, or pain medication injected next to the nerve while patients are asleep, are commonly used for pain management after shoulder surgery and are considered highly effective in decreasing post-operative pain. There are several different ways to give a nerve block. All are effective and safe. The purpose of this research is to determine if one of the available ways to give a nerve block is more effective than the others.

DETAILED DESCRIPTION:
Interscalene brachial plexus blockade is commonly performed to provide relief of postoperative pain following surgical shoulder repair. This has proven to be a reliable means of reducing the required doses of intraoperative and postoperative opiates and effectively delaying postoperative pain, as well as hastening patient discharge and increasing patient satisfaction. Neural blockade has traditionally been performed prior to surgery with the hope that preemptive analgesia will most effectively abate postoperative pain. Recently, however, it has been argued that sensitization to pain can be attributed to many factors, not solely the nociceptive battery associated with incision and subsequent intraoperative events. The duration of action and effectiveness of the treatment modality thus appear play a more important role than the actual timing of the treatment delivered. The safety and efficacy of performing interscalene brachial plexus blockade under general anesthesia has recently been reported as being not only safe, but perhaps more effective than when performed in an awake patient. We propose a randomized prospective evaluation of the analgesic efficacy comparing interscalene brachial plexus blockade performed prior to surgery with interscalene brachial plexus blockade performed following the completion of of surgery in healthy ASA I and II adolescent patients undergoing unilateral shoulder reconstruction on an outpatient basis.

ELIGIBILITY:
Inclusion Criteria:

* The subject is male or female;
* The subject is of any racial and ethnic groups;
* The subject is age 10 years to 21 years (inclusive);
* The subject is scheduled for the following
* Unilateral shoulder repair under general anesthesia on an out- patient basis, and not being performed in conjunction with any other surgical procedures;
* Agreement of the surgeon for subject participation in study.
* The subject or legally authorized representative has consented to an intra- scalene block for the procedure and the consent for the block has been obtained by an clinician (MD, DO, CRNA or APN) authorized to obtain consent who is independent of the study team
* The subject is American Society of Anesthesiologists (ASA) patient classification I-II;
* The subject's legally authorized representative has given written informed consent to participate in the study and when appropriate, the subject has given assent or consent to participate.

Exclusion Criteria:

* Additional surgical procedures are being performed concurrently;
* The subject is ASA classification > II;
* The subject has pre-existing allergies to local anesthetics;
* The subject receives sedation preoperatively;
* The subject has an imminent life threatening condition that impacts the ability to obtain informed consent;
* The subject has any other condition, which in the opinion of the principal investigator, would not be suitable for participation in the study, including but not limited preexisting neuropathy.

Ages: 10 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 79 (Actual)
Dates: Start 2013-02; Primary Completion 2025-03-31 (Estimated); Study Completion 2025-03-31 (Estimated)

PRIMARY OUTCOMES:
Pain Efficacy of Nerve Blockades | 60 minutes
  The primary outcome will be the worst pain score observed in the PACU using 0 (no pain) to 10 (worst pain) verbal Numerical Rating Scale (NRS) for pain by the study staff during the first post-operative hour.

CONTACTS AND LOCATIONS:
Overall Officials: Marc Mecoli, MD, Principal Investigator — Children's Hospital Medical Center, Cincinnati
Locations (1):
- Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio, United States

REFERENCES:
- [Background] Katz J, Clarke H, Seltzer Z. Review article: Preventive analgesia: quo vadimus? Anesth Analg. 2011 Nov;113(5):1242-53. doi: 10.1213/ANE.0b013e31822c9a59. Epub 2011 Sep 30. PMID 21965352
- [Background] Lavand'homme P. From preemptive to preventive analgesia: time to reconsider the role of perioperative peripheral nerve blocks? Reg Anesth Pain Med. 2011 Jan-Feb;36(1):4-6. doi: 10.1097/AAP.0b013e31820305b8. No abstract available. PMID 21455081
- [Background] Misamore G, Webb B, McMurray S, Sallay P. A prospective analysis of interscalene brachial plexus blocks performed under general anesthesia. J Shoulder Elbow Surg. 2011 Mar;20(2):308-14. doi: 10.1016/j.jse.2010.04.043. Epub 2010 Aug 13. PMID 20708419
- [Background] Fredrickson MJ, Ball CM, Dalgleish AJ. Analgesic effectiveness of a continuous versus single-injection interscalene block for minor arthroscopic shoulder surgery. Reg Anesth Pain Med. 2010 Jan-Feb;35(1):28-33. doi: 10.1097/AAP.0b013e3181c771bd. PMID 20048655
- [Background] Hadzic A, New York School of Regional Anesthesia: Textbook of regional anesthesia and acute pain management. New York: McGraw-Hill, Medical Pub. Division; 2007
- [Background] Angelo RL. Controversies in arthroscopic shoulder surgery: arthroscopic versus open bankart repair, thermal treatment of capsular tissue, acromioplasties--are they necessary? Arthroscopy. 2003 Dec;19 Suppl 1:224-8. doi: 10.1016/j.arthro.2003.10.005. No abstract available. PMID 14673442